CLINICAL TRIAL: NCT04124380
Title: Understanding and Testing Recovery Processes for PTSD and Alcohol Use Following Sexual Assault
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Michele Bedard-Gilligan, Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00008021; R01AA027499 (NIH); 1F32AA029865-01A1 (NIH)
Record Dates: First submitted 2019-09-23; First posted 2019-10-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Alcohol; Use, Problem; Posttraumatic Stress Disorder
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Implosive Therapy; Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Imaginal Exposure First, then Alcohol Skills (Experimental): Imaginal exposure to the sexual assault memory targeting PTSD symptoms after sexual assault. After imaginal exposure, alcohol skills targeting alcohol misuse after sexual assault.
  Interventions: Behavioral: Imaginal Exposure; Behavioral: Alcohol Skills Training
- Alcohol Skills First, then Imaginal Exposure (Experimental): Alcohol skills targeting alcohol misuse after sexual assault. After alcohol skills training, imaginal exposure to the sexual assault memory targeting PTSD symptoms after sexual assault.
  Interventions: Behavioral: Imaginal Exposure; Behavioral: Alcohol Skills Training
- Supportive Counseling/Telehealth (Active Comparator): Internet-based intervention focusing on providing support.
  Interventions: Behavioral: Supportive Telehealth
- Alcohol Skills First, no additional treatment (Experimental): Alcohol skills targeting alcohol misuse after sexual assault only. No additional treatment.
  Interventions: Behavioral: Alcohol Skills Training
- Imaginal Exposure First, no additional treatment (Experimental): Imaginal exposure to the sexual assault memory targeting PTSD symptoms after sexual assault. No additional treatment.
  Interventions: Behavioral: Imaginal Exposure

INTERVENTIONS:
Behavioral: Imaginal Exposure — Six 50 min, twice weekly video telehealth sessions will be provided based on prolonged exposure therapy for PTSD. This brief intervention includes psycho-education and focuses on imaginal exposure only based on Zoellner et al., (2016).
  Arms: Alcohol Skills First, then Imaginal Exposure; Imaginal Exposure First, no additional treatment; Imaginal Exposure First, then Alcohol Skills
Behavioral: Alcohol Skills Training — Six 50 min, twice weekly video telehealth sessions will be provided based on content from the alcohol skills training program and CBT protocols. Each session includes teaching skills and practice, focusing on mitigating rewarding aspects of alcohol, addressing cravings, and increasing other natural rewards.
  Arms: Alcohol Skills First, no additional treatment; Alcohol Skills First, then Imaginal Exposure; Imaginal Exposure First, then Alcohol Skills
Behavioral: Supportive Telehealth — The supportive counseling intervention, modeled after Litz et al. (2007), will ask participants to self-monitor their experience of weekly symptoms and complete weekly online writing about daily non-trauma related concerns and hassles. Participants will talk with a therapist on the telephone twice per week.
  Arms: Supportive Counseling/Telehealth

SUMMARY:
Sexual assault can lead to devastating consequences including the development of chronic conditions including posttraumatic stress disorder (PTSD) and alcohol use disorders (AUD). Interventions delivered soon after exposure to assault can decrease the long-term negative consequences of sexual assault but existing interventions are limited in their ability to target concurrent PTSD symptoms and alcohol use and little is known about how to make best practice treatment decisions in the early period following sexual assault. A greater emphasis on transdiagnostic processes that are related to both PTSD and alcohol use, such as fear and reward systems, can elucidate mechanisms of recovery, lead to the development of more effective intervention approaches, and guide clinical decision making for patients recently exposed to sexual assault.

DETAILED DESCRIPTION:
Following sexual assault, many individuals will develop chronic problems including posttraumatic stress disorder (PTSD) and alcohol use disorders (AUD). Intervention provided soon after assault can decrease the risk of developing chronic psychopathology and associated negative consequences. Interventions that address common underlying mechanisms of PTSD and alcohol use, such as fear and reward systems, have strong potential utility as efficacious and accessible interventions for clinicians treating patients recently exposed to sexual assault. This proposal is designed to test fear and reward as crucial processes underlying recovery following sexual assault and elucidate the most efficacious treatment targets. Employing experimental tasks (safety-signal learning paradigm and probabilistic reward task) to capture baseline underlying vulnerabilities in fear and reward systems respectively will allow for exploration of how these processes impact recovery. A randomized clinical trial (N = 180) will be conducted to test efficacy of intervention approaches that target PTSD or alcohol use compared to supportive telehealth. In addition, a phased study design will allow for exploration of efficacy of primary and secondary intervention approaches to test the questions of 1) whether it is more efficacious to target PTSD or alcohol use first; and 2) whether it is necessary to target both PTSD and alcohol use to facilitate recovery or if one is sufficient. This proposal is significant in exploring transdiagnostic mechanisms implicated in recovery following sexual assault, fear and reward, and using a novel design to compare efficacy, ordering, and necessity of two distinct intervention approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Identifies as female.
2. Between the age of 18 and 65.
3. Reports a sexual assault in the last 4 weeks to 1 year.
4. Current PTSD severity of 23+ on the PSS-I-5.
5. Current heavy alcohol use (2+ heavy episodic drinking occasions [4+ drinks on one occasion] in past month).
6. Access to the internet and a device with a webcam.

Exclusion Criteria:

1. Current diagnosis of schizophrenia, delusional disorder, or organic mental disorder as defined by the DSM-5.
2. Current diagnosis of bipolar disorder, depression with psychotic features, or depression severe enough to require immediate psychiatric treatment (i.e., serious suicide risk with intent and plan).
3. Unwilling or unable to discontinue current trauma-focused psychotherapy or current substance use psychotherapy.
4. Unstable dose of psychotropic medications in the prior 3 months.
5. Ongoing intimate relationship with the perpetrator of most recent assault.
6. Current diagnosis of a severe substance use disorder according to DSM-5, other than alcohol in the last month.
7. No clear trauma memory.
8. Current higher dose use of benzodiazepines (greater than the equivalent of 4 mg of lorazepam, 2 mg alprazolam, 1.5 mg clonazepam, or 20 mg of diazepam).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals who identify as female
Enrollment: 82 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol Use Interview | Past month
  Alcohol use will be measured using the Timeline Followback Interview (TLFB) to measure frequency and quantity of drinking behavior over the past month. The TLFB is a count of total drinks per day over the last month. Higher number of drinks on the TLFB represents higher alcohol use and worse outcomes.
Alcohol Use Self-Report | Past month
  Alcohol use will be measured using the Daily Drinking Questionnaire (DDQ) to assess for self report of typical weekly drinking (quantity, frequency). The DDQ asks for an estimated number of drinks consumed on each day in a typical week over the last month. Higher estimates for number of typical drinks each day on the DDQ represents higher alcohol use and worse outcomes.
Posttraumatic Stress Disorder Severity (PTSD) Interview | Past two weeks
  PTSD symptom severity will be measured using the Posttraumatic Stress Symptoms Scale- Interview Version for DSM-5 (PSS-I-5). The PSS-I-5 is a 20 item scale, with a minimum score of 0 and a maximum score of 80; higher values represent increased PTSD symptom severity and worse outcomes.
Posttraumatic Stress Disorder Severity (PTSD) Self-Report | Past two weeks
  PTSD symptom severity will be measured using the Posttraumatic Stress Symptoms Scale- Self-report Version for DSM-5 (PSS-SR-5). The PSS-SR-5 is a 20 item scale, with a minimum score of 0 and a maximum score of 80; higher values represent increased PTSD symptom severity and worse outcomes.

SECONDARY OUTCOMES:
Psychosocial Functioning | Past two weeks
  The single-item Global Psychosocial Functioning (GPF) item will be used as an indicator of functioning. The GPF will be reworded so as to be disorder non-specific. It is rated on a scale from 0 - 100 with higher scores representing better outcomes.
Quality of Life Functioning | Past two weeks
  The single-item Global Quality of Life (GQL) item will be used as an indicator of functioning. It is rated on a scale from 0 - 100 with higher scores representing better outcomes.
Alcohol Cravings | Past week
  The 5-item Penn Alcohol Craving Scale (PACS) will be given to assess current urges and cravings to drink alcohol. Items assess frequency, intensity, and duration of thoughts about drinking and participants rate their perceived ability to resist drinking. Total sum score on this measure ranges from 0 to 30. Higher scores represent more alcohol cravings and worse outcomes.
Alcohol Consequences | Past week
  The Short Inventory of Problems (SIP) will be given to assess alcohol related negative consequences. The SIP is a 15 item scale, with 3 items per subscale. This measure was adapted to use a time frame of the past week for responses. This measure has a minimum score of 0 and a maximum score of 15. Higher values represent increased alcohol-related problems and worse outcomes.
Depression Self-Report | Past week
  Depression will be measured with the Quick Inventory of Depressive Symptoms (QIDS-SR16) self report version. The QIDS-SR16 is a 16 item scale, with a minimum score of 0 and a maximum score of 48; higher values represent increased depression and worse outcomes.
Depression Interview | Past week
  Depression will be measured with the Quick Inventory of Depressive Symptoms (QIDS-C16) interview version. The QIDS-C16 is a 16 item scale, with a minimum score of 0 and a maximum score of 27; higher values represent increased depression and worse outcomes.
Reward | Past week
  Reward functioning will be measured with the Snaith-Hamilton Pleasure Scale (SHAPS), self-report. The SHAPS is a 14 item scale, with a minimum score of 0 and a maximum score of 14; higher values represent increased anhedonia and worse outcomes.
Fear | Past week
  Fear will be measured with the Posttrauma Avoidance Behavior Questionnaire (PABQ), self-report. The PABQ is a 25 item scale, with a minimum score of 25 and a maximum score of 100; higher values represent increased fear and worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Bedard-Gilligan, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Doherty L, Whelan M, Carter GJ, Brown K, Tarzia L, Hegarty K, Feder G, Brown SJ. Psychosocial interventions for survivors of rape and sexual assault experienced during adulthood. Cochrane Database Syst Rev. 2023 Oct 5;10(10):CD013456. doi: 10.1002/14651858.CD013456.pub2. PMID 37795783

DOCUMENTS (2):
  • Study Protocol (2019-09-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT04124380/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT04124380/SAP_001.pdf